CLINICAL TRIAL: NCT07368543
Title: Sequencing Sacituzumab Govitecan vs. Trastuzumab Deruxtecan in HER2-LOw/TROP2-High Metastatic Breast Cancer: A Randomized Phase II Study
Brief Title: Sequencing SG vs. T-DXd in HER2-Low/TROP2-High Metastatic Breast Cancer
Acronym: STORM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Director of Phase I Clinical Trial Department; Professor, Chief physician of oncology department, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2510331-4
Record Dates: First submitted 2026-01-14; First posted 2026-01-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan; trastuzumab deruxtecan

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Triple-Negative Breast Cancer) (Experimental): Patients with HER2 IHC 1+ metastatic triple-negative breast cancer (TNBC);
  Interventions: Drug: Sacituzumab Govitecan; Drug: Trastuzumab Deruxtecan
- Cohort B (HR+/HER2 IHC 1+ and Ultralow Metastatic Breast Cancer) (Experimental): Patients with HR-positive/HER2 IHC 1+ and HER2 ultralow metastatic breast cancer (MBC) who have failed endocrine therapy.
  Interventions: Drug: Sacituzumab Govitecan; Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Recommended Dose: 10 mg/kg administered by intravenous infusion on Days 1 and 8 of each 21-day treatment cycle. Continue treatment until disease progression or unacceptable toxicity.
Drug: Trastuzumab Deruxtecan — Dosage and Administration: The recommended dose is 5.4 mg/kg administered by intravenous infusion once every 3 weeks (21-day cycles). Continue treatment until disease progression or unacceptable toxicity.

SUMMARY:
Currently, no phase III RCT has directly compared SG and T-DXd sequencing strategies, and the predictive role of biomarkers remains unclear. Additionally, there is no standard scoring system for Trop-2 expression. The ASCENT trial utilized an H-score method (H-score = 3×%IHC3+ + 2×%IHC2+ + 1×%IHC1+), with scores <100, 100-200, and >200 defining low, medium, and high Trop-2 expression, respectively.This prospective study aims to: 1) Evaluate the efficacy of SG vs. T-DXd in HER2-low/Trop-2-high metastatic breast cancer, prioritizing SG for Trop-2-high patients and T-DXd for others. 2) Compare sequential treatment outcomes-T-DXd after SG failure versus SG after T-DXd failure-to inform ADC sequencing in HER2-low disease. Up to one intervening therapy is allowed before sequencing. 3) Identify biomarkers of ADC efficacy and resistance through quantitative protein analysis to optimize patient selection.

DETAILED DESCRIPTION:
This investigator-initiated study aims to evaluate the efficacy of sequential treatment with sacituzumab govitecan (SG) and trastuzumab deruxtecan (T-DXd) in patients with HER2 IHC 1+ /Trop-2-high metastatic breast cancer. It will also explore the correlation between changes in tumor-associated protein expression levels and ADC efficacy, and investigate mechanisms of ADC resistance.

The study will establish a multicenter cohort of patients treated with SG/T-DXd:

Cohort A (Triple-Negative Breast Cancer, TNBC): Includes patients with unresectable locally advanced or metastatic triple-negative breast cancer (HER2 IHC 1+) who have received ≥1 prior line of systemic therapy for metastatic disease. Prior to enrollment, all patients will undergo Trop-2 expression testing. Patients identified as Trop-2-high will be randomized 1:1 to either:SG Treatment (Trop-2 Group), orT-DXd Treatment (HER2 Group). The initially administered ADC is designated as ADC1. Upon disease progression, patients may cross over to receive the other ADC as sequential therapy (designated as ADC2). One intervening non-ADC therapy (e.g., targeted therapy, chemotherapy) is permitted prior to cross-over. Randomization will maintain a 1:1 allocation between the Trop-2 and HER2 groups.

Cohort B (HR+/HER2-ultralow or HER2 IHC 1+ Breast Cancer): Includes patients with unresectable locally advanced or metastatic HR+/HER2-ultralow or HER2 IHC 1+ breast cancer who have progressed on prior endocrine therapy. Prior to enrollment, all patients will undergo Trop-2 expression testing. Patients identified as Trop-2-high will be randomized 1:1 to either:SG Treatment (Trop-2 Group), orT-DXd Treatment (HER2 Group).

Upon progression, patients may cross over to receive the other ADC as sequential therapy. One intervening non-ADC therapy (e.g., targeted therapy, chemotherapy) is permitted prior to cross-over. Randomization will maintain a 1:1 allocation between the Trop-2 and HER2 groups.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are eligible for inclusion in this study:

* Male or female, age ≥18 years.
* ECOG performance status ≤2, with an estimated life expectancy of >3 months.
* Histologically confirmed unresectable or metastatic breast cancer that is:HER2 IHC 1+ triple-negative breast cancer, or HR-positive/HER2-ultralow or HER2 IHC 1+ breast cancer.
* Planned to receive monotherapy with Sacituzumab Govitecan and Trastuzumab Deruxtecan.
* For triple-negative breast cancer: prior systemic therapy lines ≥1.
* For HR-positive/HER2-negative metastatic breast cancer: prior endocrine therapy is required. Prior chemotherapy, immunotherapy, or targeted therapy is allowed; 0-2 lines of chemotherapy in the advanced/metastatic setting are permitted.
* Prior treatment-related adverse events have recovered to ≤Grade 1 per NCI CTCAE v5.0 (except for alopecia, non-clinically significant or asymptomatic laboratory abnormalities).
* Presence of at least one measurable or evaluable lesion.
* Willingness to provide archival or fresh tumor tissue samples for multi-omics analysis, including:

  * Baseline prior to ADC1 treatment,
  * After 2 cycles of ADC1 therapy,
  * At progression on ADC1 therapy or baseline prior to ADC2 therapy,
  * At progression on ADC2 therapy.
* FFPE tissue blocks are preferred over unstained slides. Patients must consent to tumor biopsy; if tissue is unavailable, biopsy is not feasible, or the patient declines biopsy, eligibility may be discussed and approved by the investigator.
* No severe cardiac dysfunction, with left ventricular ejection fraction (LVEF) ≥50% within 28 days before treatment.
* Adequate organ function within 7 days prior to treatment initiation:

  * Bone marrow: absolute neutrophil count (ANC) ≥1.5 × 10⁹/L; platelet count ≥100 × 10⁹/L; hemoglobin ≥90 g/L (no transfusion or blood component use within 14 days before first dose; no growth factor support within 7 days before first dose).
  * Liver: total bilirubin ≤1.5 × ULN (or <3 × ULN if Gilbert's syndrome or documented liver metastases present); ALT and AST ≤2.5 × ULN (≤5 × ULN if liver metastases present).
  * Renal: serum creatinine ≤1.5 × ULN OR creatinine clearance ≥50 mL/min (calculated by Cockcroft-Gault formula).
  * Coagulation: INR ≤1.5 × ULN and aPTT ≤1.5 × ULN (unless therapeutically anticoagulated).
* Voluntarily signed informed consent form and willingness to comply with the study protocol.
* Willingness to provide complete clinical medical record data.

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded from the study:

* Contraindication or known hypersensitivity to sacituzumab govitecan, trastuzumab deruxtecan, or any of their components (including topoisomerase I inhibitors).
* Prior treatment with sacituzumab govitecan, trastuzumab deruxtecan, or any other drug targeting the same molecular pathway.
* History of another primary malignancy, except for:

  * Malignancy treated with curative intent with no evidence of active disease for ≥2 years prior to study intervention and with low risk of recurrence, or
  * Adequately treated carcinoma in situ of the cervix, stage I endometrioid carcinoma of the uterus, or non-melanoma skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma).
* Active infection or uncontrolled systemic disease, including but not limited to:

  * Active HIV, HBV, or HCV infection,
  * Active autoimmune disease,
  * Symptomatic pleural effusion, ascites, or pericardial effusion requiring drainage,
  * Severe or uncontrolled cardiac disease requiring treatment,
  * Poorly controlled diabetes or hypertension despite medical therapy.
* Participation in another investigational drug trial within 4 weeks prior to the first study treatment (observational studies are permitted) or major surgery within 4 weeks prior to the first study treatment.
* Prior anticancer therapy within specified timeframes:

  * Chemotherapy, radiotherapy, targeted therapy, or immunotherapy within 4 weeks before the first study treatment,
  * Anticancer endocrine therapy or traditional Chinese medicine with antitumor intent within 2 weeks before the first study treatment.
* History of or current interstitial lung disease, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, or other clinically significant pulmonary disorders.
* Pregnant or breastfeeding women, or women of childbearing potential with a positive pregnancy test at baseline; patients (male or female) who are unwilling to use effective contraception throughout the study period.
* Known neurological or psychiatric disorders (e.g., epilepsy, dementia) or cognitive impairment that would compromise understanding of the study objectives, compliance, or ability to provide informed consent; or significant peripheral neuropathy.
* Primary central nervous system (CNS) tumor or untreated/symptomatic CNS metastases. Patients with asymptomatic, stable CNS metastases not requiring steroids or specific CNS-directed therapy for at least 4 weeks prior to screening may be eligible.
* Any other condition deemed unsuitable for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival 1 (PFS1) | Until progression, assessed up to approximately 24 months
  Progression-Free Survival 1 (PFS1):Time from the initiation of the first ADC (ADC1) therapy to the first occurrence of disease progression (PD) or death from any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Progression-Free Survival 2 (PFS2) | Until progression, assessed up to approximately 24 months
  Progression-Free Survival 2 (PFS2): Time from initiation of the second ADC (ADC2) therapy to the first occurrence of disease progression (PD) or death from any cause, whichever occurs earlier.
Objective Response Rate (ORR1, ORR2) | Until progression, assessed up to approximately 24 months
  Objective Response Rate (ORR1, ORR2): Proportion of patients with best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1 criteria.
Disease Control Rate (DCR | Baseline through end of study, assessed up to 24 months]
  Disease Control Rate (DCR): Proportion of patients with best overall response of CR, PR, or stable disease (SD) according to RECIST 1.1 criteria.
Overall Survival (OS) | Until death, assessed up to approximately 24 months
  Overall Survival (OS): Time from treatment initiation to death from any cause.
Safety Endpoints | Up to follow-up period, approximately 24 months]
  Safety Endpoints: Include adverse event profiles, incidence rates, dose reductions, treatment delays, and discontinuations due to adverse events.